CLINICAL TRIAL: NCT03229356
Title: An EPIC Based BPA to Enhance Quit Line Referral and Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Maryland Department of Health and Mental Hygiene (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00124880
Record Dates: First submitted 2017-07-11; First posted 2017-07-25 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Waitlist Control (No Intervention): BPA will be rolled out to waitlist control sites after 6 months
- Best Practices Advisory (BPA) (Active Comparator): Clinicians will receive an email describing the BPA and order set, along with internet links to MD Quit Line without additional supplemental education.
  Interventions: Other: Best Practices Advisory (BPA)
- BPA+ Enhanced Education (Active Comparator): Clinicians will receive an email describing the new smoking BPA, educational materials offered, and a small tutorial on using the BPA and a new smoking cessation smart set in Epic. Education materials will include the educational hand out and academic detailing from Maryland Quit Line counselors.
  Interventions: Other: BPA + Enhanced Education

INTERVENTIONS:
Other: Best Practices Advisory (BPA) — 1. BPA: The BPA is an Epic prompt that fires when a provider opens an encounter with a patient who is actively smoking. Providers will be asked to assess smoking cessation readiness and to refer patients to the free Maryland Quit Line if the patient is receptive. The Quit Line will receive an electronic referral with the patient's details. A Quit Line certified smoking cessation counselor will then call the patient at a later date and provide counseling. Receptive patient will receive up to four calls. They will receive counseling from a trained quit coach and be offered free access to NRT.
  2. Quit Line: This free telephone-based counseling service is offered to smoker in Maryland. Services offered include on-the-phone smoking cessation counseling and free nicotine replacement.
  Arms: Best Practices Advisory (BPA)
Other: BPA + Enhanced Education — BPA with Quitline Referral plus 1)Consolidated educational hand out: The hand out will include a information about counseling, pharmacotherapy, and cessation referrals 2)Online modules: Providers will be directed to optional, self-paced educational modules through the Maryland HABITS program 3)Academic detailing: This will include a single session during a clinic day in which counseling experts from the MD Quit Line will visit providers in their practice setting.
  Arms: BPA+ Enhanced Education

SUMMARY:
Smoking is the number one cause of preventable death in the United States. Given the magnitude of the problem, interventions aimed at promoting smoking cessation have the potential to make large changes in improving health outcomes. Resources to aid with smoking cessation such as telephone-based counseling are generally underutilized. The electronic medical record (EMR) in use at Johns Hopkins has limited decision support to promote referral to the Maryland Quit Line, a free smoking cessation counseling resource. The investigators propose a cluster randomized trial (Implementation-RCT hybrid design) with a waitlist control at the 22 Johns Hopkins Community Physicians (JHCP) sites, which offer primary care. The intervention will include a multi-modality intervention to promote provider use of smoking cessation resources which include an Epic-based Best Practice Advisory (BPA) that allows providers to electronically refer to the Maryland State Quit Line, educational materials, and provider visits with Quit Line representatives to review use of smoking cessation practices. Sites will be randomized to one of three arms with increasing support: 1) six-month waitlist control; 2) BPA with optional educational modules; 3) BPA with online educational modules, a quick-reference educational document, and additional visit with Quit Line representatives. The investigators hypothesize that by implementing a new Epic BPA that allows providers to easily refer to the Maryland Quit Line electronically, investigators will increase use of this resource. The investigators also hypothesize that adding additional educational materials and having Quit Line representatives perform educational outreach visits will further increase use of the Quit Line and will increase prescription of medications to assist with smoking cessation. Ultimately The investigators hope to improve patient care by increasing providers' use the Maryland Quit Line and pharmacotherapy. The investigators hope that the use of these resources will decrease smoking rates and thereby improve patient health and outcomes while improving JHCP quality metrics.

DETAILED DESCRIPTION:
Smoking is the number one cause of preventable death in the United States. Given the magnitude of the problem, interventions aimed at promoting smoking cessation have the potential to make large changes in improving health outcomes. Resources to aid with smoking cessation such as telephone-based counseling are generally underutilized. The electronic medical record (EMR) in use at Johns Hopkins has limited decision support to promote referral to the Maryland Quit Line, a free smoking cessation counseling resource. The investigators propose a cluster randomized trial (Implementation-RCT hybrid design) with a waitlist control at the 22 Johns Hopkins Community Physicians (JHCP) sites, which offer primary care. The intervention will include a multi-modality intervention to promote provider use of smoking cessation resources which include an Epic-based Best Practice Advisory (BPA) that allows providers to electronically refer to the Maryland State Quit Line, educational materials, and provider visits with Quit Line representatives to review use of smoking cessation practices. Sites will be randomized to one of three arms with increasing support: 1) six-month waitlist control; 2) BPA with optional educational modules; 3) BPA with online educational modules, a quick-reference educational document, and additional visit with Quit Line representatives. The investigators hypothesize that by implementing a new Epic BPA that allows providers to easily refer to the Maryland Quit Line electronically, The investigators will increase use of this resource. The investigators also hypothesize that adding additional educational materials and having Quit Line representatives perform educational outreach visits will further increase use of the Quit Line and will increase prescription of medications to assist with smoking cessation. Ultimately, the investigators hope to improve patient care by increasing providers' use the Maryland Quit Line and pharmacotherapy. The investigators hope that the use of these resources will decrease smoking rates and thereby improve patient health and outcomes while improving JHCP quality metrics.

The primary goal of this study is to test the effectiveness of instituting an Epic BPA in increasing Maryland Quit Line referrals. The secondary goals are to measure the BPA's effect and the effect of additional provider education on patient engagement with the Quit Line, and on prescription of medications that aid in smoking cessation.

Aim 1: In a three-arm, cluster randomized trial, to test the effectiveness of an Epic BPA with provider educational support and provider detailing in provision of smoking cessation services.

Hypothesis 1: An Epic-based BPA to prompt providers to electronically refer people who are ready to quit smoking to the Maryland Quit Line will increase use of this service compared to waitlist control.

Hypothesis 2: An Epic-based BPA supplemented with educational materials and academic detailing will increase Quit-Line referral compared to control.

Hypothesis 3: Additional provider support including educational materials, in-person academic detailing, will increase successful referrals to the Quit Line and prescription of cessation pharmacotherapy compared to waitlist control and BPA only

ELIGIBILITY:
Inclusion Criteria:

* Johns Hopkins Community Physicians Primary Care Practices (Internal Medicine and Family Medicine)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geetanjali Chander, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Community Physcians, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu SS, Neff L, Agaku IT, Cox S, Day HR, Holder-Hayes E, King BA. Tobacco Product Use Among Adults - United States, 2013-2014. MMWR Morb Mortal Wkly Rep. 2016 Jul 15;65(27):685-91. doi: 10.15585/mmwr.mm6527a1. PMID 27416365
- [Background] Stead LF, Hartmann-Boyce J, Perera R, Lancaster T. Telephone counselling for smoking cessation. Cochrane Database Syst Rev. 2013 Aug 12;(8):CD002850. doi: 10.1002/14651858.CD002850.pub3. PMID 23934971
- [Background] Sharifi M, Adams WG, Winickoff JP, Guo J, Reid M, Boynton-Jarrett R. Enhancing the electronic health record to increase counseling and quit-line referral for parents who smoke. Acad Pediatr. 2014 Sep-Oct;14(5):478-84. doi: 10.1016/j.acap.2014.03.017. PMID 25169159
- [Background] Bernstein SL, Weiss J, DeWitt M, Tetrault JM, Hsiao AL, Dziura J, Sussman S, Miller T, Carpenter K, O'Connor P, Toll B. A randomized trial of decision support for tobacco dependence treatment in an inpatient electronic medical record: clinical results. Implement Sci. 2019 Jan 22;14(1):8. doi: 10.1186/s13012-019-0856-8. PMID 30670043
- [Background] Boyle R, Solberg L, Fiore M. Use of electronic health records to support smoking cessation. Cochrane Database Syst Rev. 2014 Dec 30;2014(12):CD008743. doi: 10.1002/14651858.CD008743.pub3. PMID 25547090
- [Background] Carson KV, Verbiest ME, Crone MR, Brinn MP, Esterman AJ, Assendelft WJ, Smith BJ. Training health professionals in smoking cessation. Cochrane Database Syst Rev. 2012 May 16;2012(5):CD000214. doi: 10.1002/14651858.CD000214.pub2. PMID 22592671
- [Background] O'Brien MA, Rogers S, Jamtvedt G, Oxman AD, Odgaard-Jensen J, Kristoffersen DT, Forsetlund L, Bainbridge D, Freemantle N, Davis DA, Haynes RB, Harvey EL. Educational outreach visits: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD000409. doi: 10.1002/14651858.CD000409.pub2. PMID 17943742
- [Background] Soumerai SB, Avorn J. Principles of educational outreach ('academic detailing') to improve clinical decision making. JAMA. 1990 Jan 26;263(4):549-56. PMID 2104640
- [Derived] Wadlin J, Ford DE, Albert MC, Wang NY, Chander G. Implementing an EMR-Based Referral for Smoking Quitline Services with Additional Provider Education, a Cluster-Randomized Trial. J Gen Intern Med. 2022 Aug;37(10):2438-2445. doi: 10.1007/s11606-021-07275-6. Epub 2022 Mar 8. PMID 35260960

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Waitlist Control Sites A and B were together (8) in the first 6 months after which they were randomized to A (4) and B (4).
Units Other Than Participants: Practice Sites
Groups:
- Waitlist Control - A: BPA+ Enhanced Education will be rolled out to waitlist control sites after 6 months.
- Waitlist Control - B: BPA will be rolled out to waitlist control sites after 6 months.
- Best Practices Advisory (BPA): Clinicians will receive an email describing the BPA and order set, along with internet links to MD Quit Line without additional supplemental education.
  Best Practices Advisory (BPA): 1. BPA: The BPA is an Epic prompt that fires when a provider opens an encounter with a patient who is actively smoking. Providers will be asked to assess smoking cessation readiness and to refer patients to the free Maryland Quit Line if the patient is receptive. The Quit Line will receive an electronic referral with the patient's details. A Quit Line certified smoking cessation counselor will then call the patient at a later date and provide counseling. Receptive patient will receive up to four calls. They will receive counseling from a trained quit coach and be offered free access to NRT.
  2. Quit Line: This free telephone-based counseling service is offered to smoker in Maryland. Services offered include on-the-phone smoking cessation counseling and free nicotine replacement.
Period: Phase 1 (Months 1-6)
Arm/Group | Waitlist Control - A | Waitlist Control - B | Best Practices Advisory (BPA) | BPA+ Enhanced Education
Started | NA; 4 Practice Sites (Number of participants is not available for this study, only practice-level data collected.) | NA; 4 Practice Sites (Number of participants is not available for this study, only practice-level data collected.) | NA; 7 Practice Sites (Number of participants is not available for this study, only practice-level data collected.) | NA; 7 Practice Sites (Number of participants is not available for this study, only practice-level data collected.)
Completed | NA; 4 Practice Sites (Number of participants is not available for this study, only practice-level data collected.) | NA; 4 Practice Sites (Number of participants is not available for this study, only practice-level data collected.) | NA; 7 Practice Sites (Number of participants is not available for this study, only practice-level data collected.) | NA; 7 Practice Sites (Number of participants is not available for this study, only practice-level data collected.)
Not Completed | NA; 0 Practice Sites | NA; 0 Practice Sites | NA; 0 Practice Sites | NA; 0 Practice Sites
Period: Phase 2 (Months 7-12)
Arm/Group | Waitlist Control - A | Waitlist Control - B | Best Practices Advisory (BPA) | BPA+ Enhanced Education
Started | NA; 4 Practice Sites (Number of participants is not available for this study, only practice-level data collected.) | NA; 4 Practice Sites (Number of participants is not available for this study, only practice-level data collected.) | NA; 7 Practice Sites (Number of participants is not available for this study, only practice-level data collected.) | NA; 7 Practice Sites (Number of participants is not available for this study, only practice-level data collected.)
Completed | NA; 4 Practice Sites (Number of participants is not available for this study, only practice-level data collected.) | NA; 4 Practice Sites (Number of participants is not available for this study, only practice-level data collected.) | NA; 7 Practice Sites (Number of participants is not available for this study, only practice-level data collected.) | NA; 7 Practice Sites (Number of participants is not available for this study, only practice-level data collected.)
Not Completed | NA; 0 Practice Sites | NA; 0 Practice Sites | NA; 0 Practice Sites | NA; 0 Practice Sites

BASELINE CHARACTERISTICS:
Population: Number of participants is not available for this study, only practice-level data collected.
Units Other Than Participants: Practice Sites
Groups:
- Total: Total of all reporting groups
Arm/Group | Waitlist Control - A | Waitlist Control - B | Best Practices Advisory (BPA) | BPA+ Enhanced Education | Total
Number analyzed (Participants) | NA | NA | NA | NA | NA
Number analyzed (Practice Sites) | 4 | 4 | 7 | 7 | 22
Age, Customized [Number; unit: participants] — No age data was collected.
Sex/Gender, Customized [Number; unit: participants] — No sex data was collected.
Race/Ethnicity, Customized [Number; unit: participants] — Race/Ethnicity data was not collected.
Region of Enrollment [Number; unit: Practice Sites]
  United States | 4 | 4 | 7 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: Provider Electronic Referrals to the Maryland Quit Line
Description: Number of referrals made out of total eligible for referral.
Time Frame: 6 months
Population: This assessment was on number of service referrals made out of eligible encounters and not individual participants. Individual participants analyzed was not collected. Referrals were not made for Waitlist control groups A and B because they were not randomized yet at this time to either BPA or BPA+ Enhanced Education. Data not collected from the waitlist groups at this time point as the intervention had not been rolled out.
Measure: Number; unit: referrals
Units Other Than Participants: Eligible Encounters
Arm/Group | Waitlist Control - A | Waitlist Control - B | Best Practices Advisory (BPA) | BPA+ Enhanced Education
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (Eligible Encounters) | 0 | 0 | 6857 | 5636
referrals |  |  | 623 | 405

2. Secondary Outcome: Prescription of Pharmacotherapy for Smoking Cessation
Description: Nicotine replacement, Varenicline or Bupropion prescription.
Time Frame: 12 months
Population: Data was not collected for this outcome measure.
Arm/Group | Waitlist Control - A | Waitlist Control - B | Best Practices Advisory (BPA) | BPA+ Enhanced Education
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Patient Engagement With the Quit Line
Description: Number of patients that accepted services or declined or were not reached or were already enrolled.
Time Frame: 6 months
Population: This assessment was on number of service referrals and not individual participants. Individual participants analyzed was not collected. This assessment was not done for Waitlist control groups A and B. Due to differences in the timeline of data collection between data from the EMR (within the trial period) and those received from the quitline (monthly summary reports), there are minor discrepancies between the referral totals of this outcome and outcome 1.
Measure: Number; unit: service referrals
Units Other Than Participants: Number of service referrals
Arm/Group | Waitlist Control - A | Waitlist Control - B | Best Practices Advisory (BPA) | BPA+ Enhanced Education
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (Number of service referrals) | 0 | 0 | 626 | 392
service referrals
  Accepted services |  |  | 133 | 80
  Declined |  |  | 27 | 17
  Already enrolled |  |  | 6 | 4
  Not reached |  |  | 346 | 216
  Pending/incomplete |  |  | 114 | 75

4. Secondary Outcome: Provider Electronic Referrals to the Maryland Quit Line
Description: Number of referrals made out of total eligible for referral.
Time Frame: 12 months
Population: This assessment was on number of service referrals made out of eligible encounters and not individual participants. Individual participants analyzed was not collected.
Measure: Number; unit: referrals
Units Other Than Participants: Eligible Encounters
Arm/Group | Waitlist Control - A | Waitlist Control - B | Best Practices Advisory (BPA) | BPA+ Enhanced Education
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (Eligible Encounters) | 3635 | 3337 | 5797 | 4881
referrals | 272 | 186 | 284 | 203

5. Secondary Outcome: Patient Engagement With the Quit Line
Description: Number of patients that accepted services or declined or were not reached or were already enrolled.
Time Frame: 12 months
Population: This assessment was on number of service referrals and not individual participants. Individual participants analyzed was not collected. This assessment was not done for Waitlist control groups A and B.
Measure: Number; unit: service referrals
Units Other Than Participants: Number of service referrals
Arm/Group | Waitlist Control - A | Waitlist Control - B | Best Practices Advisory (BPA) | BPA+ Enhanced Education
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (Number of service referrals) | 0 | 0 | 514 | 487
service referrals
  Accepted services |  |  | 100 | 80
  Declined |  |  | 80 | 77
  Already enrolled |  |  | 6 | 7
  Not reached |  |  | 289 | 291
  Pending/incomplete |  |  | 39 | 32

ADVERSE EVENTS:
Description: Adverse events were not assessed.
Arm/Group | Waitlist Control - A | Waitlist Control - B | Best Practices Advisory (BPA) | BPA+ Enhanced Education
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT03229356/Prot_SAP_000.pdf